CLINICAL TRIAL: NCT07013669
Title: Receptive Music Interventions During Intradermal Testing in Children: A Randomized Controlled Trial Comparing Solfeggio Frequencies and Turkish Classical Music on Pain and Parental Anxiety
Brief Title: Receptive Music Interventions During Intradermal Testing in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Gungor (Other)
Responsible Party: Sponsor-Investigator, Hilal Gungor, Medical Doctor, Pediatric Allergy and Immunology, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-276166482
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Music Therapy; Anxiety; Pain Management; Skin Tests; Child
MeSH Terms: conditions — Anxiety Disorders; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants undergo standard intradermal testing (IDT) without any additional auditory intervention
- Solfeggio Music Intervention (Experimental): Participants receive receptive music therapy using Solfeggio frequencies (174 Hz, 285 Hz, 396 Hz, and 528 Hz) during the IDT procedure. Music starts five minutes before and continues throughout the procedure
  Interventions: Behavioral: Receptive Music Therapy - Solfeggio Frequencies
- Traditional Turkish Music Intervention (Experimental): Participants receive receptive music therapy using selected Traditional Turkish Music modes (makams), including Rast, Hicaz, Uşşak, Neva, and Saba, during the IDT procedure. Music starts five minutes before and continues throughout the procedure
  Interventions: Behavioral: Receptive Music Therapy - Traditional Turkish Music

INTERVENTIONS:
Behavioral: Receptive Music Therapy - Solfeggio Frequencies — Music featuring Solfeggio frequencies (174 Hz, 285 Hz, 396 Hz, 528 Hz) is played through standardized speakers in a sound-isolated room during IDT. Duration includes five minutes before and throughout the procedure
  Arms: Solfeggio Music Intervention
Behavioral: Receptive Music Therapy - Traditional Turkish Music — Selected Turkish Classical Music pieces (makams: Rast, Hicaz, Uşşak, Neva, Saba) are played via speakers in a sound-isolated room during IDT. Music begins five minutes prior and continues during the procedure.
  Arms: Traditional Turkish Music Intervention

SUMMARY:
The study summary and design were to assess procedural anxiety and stress in parents and pain perception in children during intradermal testing. Music medicine was incorporated into the study design as a nonpharmacological intervention. Two distinct auditory modalities were used: solfeggio frequencies-174 Hz, 285 Hz, 396 Hz, and 528 Hz-which have been suggested to interact with the human energy field through resonance-based mechanisms, and Turkish classical musical modes (makams), such as Rast, Hicaz, Uşşak, Neva, and Saba, which are modal systems that include microtonal intervals and follow specific melodic progressions that are often associated with different emotional and spiritual effects as well as sensory and emotional regulation potential.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 2 and 17 years
2. Referred to the Pediatric Allergy Clinic for evaluation of suspected drug hypersensitivity reactions
3. Accompanied by a parent or legal guardian willing to participate
4. Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

1. Known neurological, psychiatric, or developmental disorders in the child
2. Use of sedatives or analgesic medications within 24 hours prior to testing
3. Hearing impairment or auditory processing disorders in the child4.Non-consent or withdrawal of consent by parent or guardian
4. Inability of the parent to complete anxiety assessments (e.g., due to language or cognitive barriers)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change in Parental State Anxiety Levels | within 5 minutes before and post procedure
  Change in parental state anxiety will be assessed using the State-Trait Anxiety Inventory - State Subscale (STAI-S). The STAI-S is a validated psychological inventory that measures current levels of anxiety. It consists of 20 items, each rated on a 4-point Likert scale, with total scores ranging from 20 to 80. Higher scores indicate greater levels of anxiety.
  STAI-S scores will be collected immediately before and immediately after the intradermal testing (IDT) procedure. The change in anxiety levels will be calculated as the difference between post-procedure and pre-procedure scores (ΔSTAI-S), and will be used to evaluate the effect of the intervention.
Pain Levels in Pediatric Patients During Intradermal Testing | within 2 minutes post-procedure
  Pain scores will be evaluated immediately after the intradermal testing (IDT) procedure.
  For children under 5 years of age, pain will be assessed using the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS). This is a behavioral pain assessment tool with scores ranging from 4 to 13, where higher scores indicate greater pain.
  For children aged 5 years and older, pain will be assessed using the Wong-Baker FACES Pain Rating Scale. This self-report scale ranges from 0 to 10, where higher scores indicate greater pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof Dr Cemil Tascioglu Education and Research Hospital Organization, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Identified individual participant data (IPD) that underlie the results reported in this article will be shared. This includes:Demographic information (age, sex, parental education level)Baseline clinical data (allergy history, suspected drug, clinical symptoms)Pre- and post-intervention STAI scores (State and Trait Anxiety Inventory)Pain scores measured using CHEOPS and Wong-Baker FACES scalesGroup allocation (Control, Solfeggio, Traditional Turkish Music)All shared data will be anonymized to protect participant confidentiality.
Supporting Information: Study Protocol